CLINICAL TRIAL: NCT04977258
Title: Effect of Different Hydration Strategies on Autonomic Acceleration During Recovery in Individuals With Coronary Artery Disease Undergoing Aerobic Exercise
Brief Title: Different Hydration Strategies Associated With Aerobic Exercise In Coronary
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Responsible Party: Principal Investigator, Luiz Carlos Marques Vanderlei, Principal Investigator, Universidade Estadual Paulista Júlio de Mesquita Filho
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 34722320.0.0000.5402
Record Dates: First submitted 2021-07-15; First posted 2021-07-26 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-08

CONDITIONS: Coronary Disease
Keywords: Autonomic Nervous System; Fluid Therapy; Heart Rate; Exercise
MeSH Terms: conditions — Coronary Disease; Motor Activity | interventions — Drinking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Active Comparator): Only treadmill aerobic exercise with 60 min recovery in supine position.
  Interventions: Other: Treadmill aerobic exercise without water intake
- Controlled hydration group (Experimental): Treadmill aerobic exercise with 60 min recovery in supine position, with mineral water predetermined intake.
  Interventions: Other: Treadmill aerobic exercise with water intake of a predetermined amount.
- Ad Libitum hydration group (Experimental): Treadmill aerobic exercise with 60 min recovery in supine position, with mineral water intake in an uncontrolled manner.
  Interventions: Other: Treadmill aerobic exercise with water intake according to the desire to drink

INTERVENTIONS:
Other: Treadmill aerobic exercise without water intake — The volunteers will be submitted to a cardiovascular rehabilitation session with 40 minutes of treadmill aerobic exercise followed by 60 minutes of recovery at the supine position.
  Arms: Control group
Other: Treadmill aerobic exercise with water intake of a predetermined amount. — The volunteers will be submitted to a cardiovascular rehabilitation session with 40 minutes of treadmill aerobic exercise and water intake followed by 60 minutes of recovery at the supine position.
  Arms: Controlled hydration group
Other: Treadmill aerobic exercise with water intake according to the desire to drink — The volunteers will be submitted to a cardiovascular rehabilitation session with 40 minutes of treadmill aerobic exercise and water intake followed by 60 minutes of recovery at the supine position.
  Arms: Ad Libitum hydration group

SUMMARY:
The need to restore water losses resulting from physical activity has become established and diffused into international consensus for healthy individuals or high-performance athletes. However, the influence of fluid replacement when administered during and after exercise on cardiac autonomic modulation with autonomic alterations known as the coronary arteries remain poorly understood. The aim of the study was to evaluate and compare whether different hydration strategies are able to promote acceleration of the recovery of autonomic modulation in individuals with coronary artery disease undergoing aerobic exercise. This study is a cross-over clinical trial, which will be developed based on an experimental procedure performed in four stages. A total of 31 individuals will be recruited in this study and will perform four standardized cardiovascular rehabilitation (CR) sessions. The participants will perform CR with mineral water intake in phase three and four. In phase three, the consumption will be done a quantity of water predetermined by the evaluator, based on the loss of body mass measured in the second session. In phase four, hydration will be carried out in an uncontrolled manner, according to the desire to drink water during the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Men with coronary heart disease ischemia, over 45 years
* At least three months of cardiovascular rehabilitation

Exclusion Criteria:

* Smokers, alcoholics
* Uncontrolled metabolic disease (eg, uncontrolled diabetes and thyroid diseases)
* Abnormal hemodynamic responses during exercise such as disproportionate increase / fall of heart rate and / or blood pressure to low / high levels of load
* Myocardial ischemia and / or severe ventricular arrhythmias during the exercise test

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2021-08-16 (Estimated); Primary Completion 2021-10-26 (Estimated); Study Completion 2022-02-26 (Estimated)

PRIMARY OUTCOMES:
Heart rate variability | up to six months
  Linear indices of heart rate variability in the time domain (SDNN, rMSSD).
Heart rate variability | up to six months
  Linear indices of heart rate variability in the frequency domain (HF, LF, LF/HF)
Heart rate variability | up to six months
  Geometric indices of heart rate variability (TINN, RRTRI, SD1, SD2, SD1/SD2)

CONTACTS AND LOCATIONS:
Overall Officials: Luiz Carlos Vanderlei, PhD, Study Director — Universidade Estadual Paulista - UNESP - Campus de Presidente Prudente
Locations (1):
- Luiz Carlos Masques Vanderlei, Presidente Prudente, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No